CLINICAL TRIAL: NCT00759408
Title: The Role of Endothelin in Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anju Nohria, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999-P-003126
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Hypertension
Keywords: primary pulmonary hypertension; secondary pulmonary hypertension due to left heart failure; secondary pulmonary hypertension due to other causes; patients without pulmonary disease or pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension | interventions — cyclo(Trp-Asp-Pro-Val-Leu)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): BQ-123
  Interventions: Drug: BQ-123

INTERVENTIONS:
Drug: BQ-123 — 6-120 µg/min

SUMMARY:
The purpose of the study is is to determine the effect, on the lung circulation, of BQ-123, an investigational compound which is not approved by the FDA.

DETAILED DESCRIPTION:
Endothelin levels are increased in patients with pulmonary hypertension. We wish to compare the effect of an endothelin antagonist on pulmonary hypertension due to a variety of causes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers or known diagnosis of pulmonary hypertension

Exclusion Criteria:

* hypertension due to other reasons (not pulmonary)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 1999-02; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Creager, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BQ-123: BQ-123 (6-120 µg/min) will be administered intravenously.
Period: Overall Study
Arm/Group | BQ-123
Started | 38
Completed | 19
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | BQ-123
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vascular Resistance (PVR)
Description: PVR will be measured at these 5 time points: 1) Baseline, 2) Hypoxia induced and maintained for 15 min post-baseline at which time the measurement is taken again, 3) Baseline oxygen saturation (Normoxia) reestablished 15 min post-hypoxia period, at which time the measurement is taken again 4) Normoxia measurement taken after BQ-123 administered for 60 min after time point 3, 5) Hypoxia induced and maintained for 15 min after BQ-123 normoxia period, at which time the measurement is taken again.
Time Frame: Baseline and time points 2, 3, 4, and 5 (as described in Outcome Measure Description)
Population: Only 19 healthy volunteers completed the study. The study was closed before the 19 patients with established pulmonary hypertension could have data collected.
Measure: Mean (Standard Error); unit: dyn*sec/cm^5
Arm/Group | BQ-123
Number analyzed (Participants) | 19
dyn*sec/cm^5
  Baseline | 64 (5)
  Time 2: Hypoxia | 119 (10)
  Time 3: Normoxia | 67 (5)
  Time 4: Normoxia/BQ-123 | 46 (5)
  Time 5: Hypoxia/BQ-123 | 85 (9)

2. Secondary Outcome: Systemic Vascular Resistance (SVR)
Description: SVR will be measured at these 5 time points: 1) Baseline, 2) Hypoxia induced and maintained for 15 min post-baseline at which time the measurement is taken again, 3) Baseline oxygen saturation (Normoxia) reestablished 15 min post-hypoxia period, at which time the measurement is taken again 4) Normoxia measurement taken after BQ-123 administered for 60 min after time point 3, 5) Hypoxia induced and maintained for 15 min after BQ-123 normoxia period, at which time the measurement is taken again.
Time Frame: Baseline and time points 2, 3, 4, and 5 (as described in Outcome Measure Description)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: dyn*sec/cm^5
Arm/Group | BQ-123
Number analyzed (Participants) | 19
dyn*sec/cm^5
  Baseline | 1368 (52)
  Time 2: Hypoxia | 1050 (57)
  Time 3: Normoxia | 1351 (44)
  Time 4: Normoxia/BQ-123 | 1069 (38)
  Time 5: Hypoxia/BQ-123 | 828 (43)

3. Secondary Outcome: Mean Pulmonary Artery Pressure (PAP)
Description: PAP will be measured at these 5 time points: 1) Baseline, 2) Hypoxia induced and maintained for 15 min post-baseline at which time the measurement is taken again, 3) Baseline oxygen saturation (Normoxia) reestablished 15 min post-hypoxia period, at which time the measurement is taken again 4) Normoxia measurement taken after BQ-123 administered for 60 min after time point 3, 5) Hypoxia induced and maintained for 15 min after BQ-123 normoxia period, at which time the measurement is taken again.
Time Frame: Baseline and time points 2, 3, 4, and 5 (as described in Outcome Measure Description)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | BQ-123
Number analyzed (Participants) | 19
mmHg
  Baseline | 10 (1)
  Time 2: Hypoxia | 15 (1)
  Time 3: Normoxia | 10 (1)
  Time 4: Normoxia/BQ-123 | 9 (1)
  Time 5: Hypoxia/BQ-123 | 14 (1)

4. Secondary Outcome: Cardiac Output (CO)
Description: CO will be measured at these 5 time points: 1) Baseline, 2) Hypoxia induced and maintained for 15 min post-baseline at which time the measurement is taken again, 3) Baseline oxygen saturation (Normoxia) reestablished 15 min post-hypoxia period, at which time the measurement is taken again 4) Normoxia measurement taken after BQ-123 administered for 60 min after time point 3, 5) Hypoxia induced and maintained for 15 min after BQ-123 normoxia period, at which time the measurement is taken again.
Time Frame: Baseline and time points 2, 3, 4, and 5 (as described in Outcome Measure Description)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: l/min
Arm/Group | BQ-123
Number analyzed (Participants) | 19
l/min
  Baseline | 5.3 (0.3)
  Time 2: Hypoxia | 6.7 (0.4)
  Time 3: Normoxia | 5.2 (0.3)
  Time 4: Normoxia/BQ-123 | 6.4 (0.3)
  Time 5: Hypoxia/BQ-123 | 8.3 (0.6)

ADVERSE EVENTS:
Arm/Group | BQ-123
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No